CLINICAL TRIAL: NCT02177838
Title: Selecting for Cetuximab Responders in Advanced Head and Neck SCC
Brief Title: Cetuximab and Radiation Therapy in Treating Patients With Stage III-IV Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Sung Kim, MD, Residency and Clinical Director, Residency & Clinical Director, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20150001420; NCI-2014-01303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 031204 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Larynx; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cetuximab, cisplatin, EBRT) (Experimental): Patients receive cetuximab IV over 60-120 minutes for 3 weeks. Patients then undergo EBRT over 6-7 weeks. Patients achieving response continue weekly doses of cetuximab until radiation therapy is completed. Patients unable to achieve response or progression receive cisplatin IV over 1-2 hours on days 1, 22, and 43 of radiation therapy.
  Interventions: Biological: cetuximab; Drug: cisplatin; Radiation: external beam radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Radiation: external beam radiation therapy — Undergo EBRT
  Other Names: EBRT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies cetuximab and radiation therapy in treating patients with stage III-IV head and neck cancer. Monoclonal antibodies, such as cetuximab, may block tumor growth in different ways by targeting certain cells. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cetuximab or cisplatin together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. 2 year (yr) locoregional control in cetuximab responders.

SECONDARY OBJECTIVES:

I. Assess secondary clinical endpoints such as the percent of patients receiving neoadjuvant cetuximab who progress by computed tomography (CT) Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria during the neoadjuvant cetuximab, the 2 yr locoregional control for non-responders to neoadjuvant cetuximab, and the complete response rate to positron emission tomography (PET)/computed tomography (CT) scan 3 months after the completion of radiation therapy for both responders and for non-responders to neoadjuvant cetuximab.

II. Analyze the relationship of known deoxyribonucleic acid (DNA) mutations in tumor per the FoundationOne genomic profile, and correlate to clinical endpoints such as locoregional control.

II. Analyze any changes in protein production at the tumor in response to 3 weeks of cetuximab.

III. Analyze any changes in protein production at the skin in response to 3 weeks of cetuximab.

IV. To investigate whether the tumor imaging characteristics including anatomical and molecular parameters evaluated by PET/CT, either alone or combined with other biomarkers can attribute to the better prediction for the clinical outcomes, as the response to neoadjuvant cetuximab; and the final clinical endpoint, the 2-year local regional controls.

OUTLINE:

Patients receive cetuximab intravenously (IV) over 60-120 minutes for 3 weeks. Patients then undergo external beam radiation therapy (EBRT) over 6-7 weeks. Patients achieving response continue weekly doses of cetuximab until radiation therapy is completed. Patients unable to achieve response or progression receive cisplatin IV over 1-2 hours on days 1, 22, and 43 of radiation therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the oropharynx, hypopharynx or larynx
* Stage III/IVa/b squamous cell carcinoma (SCC) by American Joint Committee on Cancer (AJCC) 7 criteria (advanced, but not metastatic)
* Patients must give informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Platelets >= 100,000/uL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Hemoglobin > 8 g/dl (use of transfusion to achieve this is acceptable)
* Total bilirubin < 2 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional ULN
* Serum creatinine < 2 x institutional ULN or creatinine clearance > 50 ml/min as determined by 24 hour collection or estimated by Cockcroft-Gault formula
* Estimated life expectancy of at least 12 weeks
* Negative pregnancy test

Exclusion Criteria:

* Patients may not have received previous therapy for their head and neck SCC, including chemotherapy, radiation therapy, or surgery beyond biopsy
* Second primary malignancy; exceptions are 1) patient had a second primary malignancy but has been treated and disease free for at least 3 years, 2) in situ carcinoma (e.g. in situ carcinoma of the cervix), 3) non-melanomatous carcinoma of the skin
* Patients with metastatic disease beyond the neck and supraclavicular region will be excluded
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator; this includes scleroderma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab or cisplatinum or other agents used in the study
* Women who are pregnant; women of childbearing age must agree to undergo a pregnancy test prior to therapy and to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with human immunodeficiency virus (HIV) infection are not automatically excluded, but must meet the following criteria: cluster of differentiation (CD)4 count is > 499/cu mm and their viral load is < 50 copies/ml; use of highly active anti-retroviral therapy (HAART) is allowed
* Patients who have had either myocardial infarction, coronary artery bypass graft, coronary artery stenting, hospital admission for heart related issues such as congestive heart failure or arrhythmia within the last 3 months, will not be allowed on protocol
* Grade 3-4 electrolyte abnormalities (Common Terminology Criteria for Adverse Events [CTCAE], version [v]. 4):

  * Serum calcium (ionized or adjusted for albumin) < 7 mg/dl (1.75 mmol/L) or > 12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels
  * Magnesium < 0.9 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels
  * Potassium < 3.5 mmol/L or > 6 mmol/L despite intervention to normalize levels
  * Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kim, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
Started | 8
Completed | 5
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Locoregional Control in Cetuximab Responders
Description: Target number of patients for the study was 27. At the termination of the study, 8 patients were accrued and finished treatment but 1 patient dropped out before follow up, leaving an evaluable number of 7. As the enrollment in the study did not reach the target number of patients, we were not able to produce statistically reliable results to detect the expected difference. Therefore, we have decided to provide summary statistics of primary and secondary outcomes.
  Among 3 cetuximab responders, two did not have progression within 2 year follow-up time and one had a locoregional recurrence and expired.
Time Frame: 2 years
Population: Target number of patients for the study was 27. At the termination of the study, 8 patients were accrued and finished treatment but 1 patient dropped out before follow up, leaving an evaluable number of 7. As the enrollment in the study did not reach the target number of patients, we were not able to produce statistically reliable results to detect the expected difference.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Percent of Patients Who Progress During Neoadjuvant Cetuximab by CT RECIST 1.1 Criteria
Description: Among 7 patients, no one progressed during neoadjuvant cetuximab per RECIST 1.1 CT criteria (0%).
Time Frame: Day 14-21 after the first dose of cetuximab
Population: This measure what not evaluated because the study was halted prematurely due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
Number analyzed (Participants) | 7
Participants | 0

3. Secondary Outcome: Locoregional Control for Non-responders to Neoadjuvant Cetuximab
Description: Among 4 cetuximab non-responders, none had locoregional failure at 2 years. Two patients had known HPV status; one patient was HPV+ and another patient HPV-. HPV status for the other two was unknown. HPV positive patient had no sign of progression within 2 years of follow-up. HPV negative patient had no sign of progression for 210 days until the last follow-up. One HPV unknown patient did not show progression within 2 years of follow-up, and the other HPV unknown patient had no progression for 115 days until the last follow-up.
Time Frame: 2 years
Population: This measure what not evaluated because the study was halted prematurely due to low accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: All patients who received one dose of protocol therapy were evaluated for assessment of toxicity. All adverse events, whether observed by the treating physician or reported by the patient, occurring during the active portion of therapy or up to 30 days after the last dose of treatment were captured.
Arm/Group | Treatment (Cetuximab, Cisplatin, EBRT)
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cetuximab, Cisplatin, EBRT) (N=8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cetuximab, Cisplatin, EBRT) (N=8)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
White blood cell count decreased (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 7 (7)
Dehydration (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck pain
Dysgeusia (Nervous system disorders) | 4 (4)
Pain (General disorders) | 2 (2) — Headache
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 5 (5) — Sore throat
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneform (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the trial led to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02177838/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02177838/ICF_001.pdf